CLINICAL TRIAL: NCT05856071
Title: Effects of Clamshell Exercises in Terminal Extension Lag After Anterior Cruciate Ligament
Brief Title: TEL and Clam Shell Exercises Affect After ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR /23/0119 sohaib Kaleem
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Knee Ligament Injury
Keywords: anterior cruciate ligament reconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clamshells exercises (Experimental)
  Interventions: Device: goniometer; Other: clamshells exercises
- traditional physical therapy (Active Comparator)
  Interventions: Device: goniometer; Other: traditional physical therapy

INTERVENTIONS:
Device: goniometer — to measure the range of motion
Other: clamshells exercises — clamshells exercises
  Arms: clamshells exercises
Other: traditional physical therapy — traditional physical therapy
  Arms: traditional physical therapy

SUMMARY:
The purpose of this study to determine the effects of the addition of isolated hip strengthening exercises to traditional rehabilitation after Anterior cruciate ligament reconstruction (ACLR). Clamshells exercises unique in scene because it mainly focuses on the muscle surrounding the hip whereas the traditional exercises mostly paid attention on quads and hams exercise

DETAILED DESCRIPTION:
In 2020, researcher conducted a randomized controlled clinical trial to determine "Does six-weeks of Hip-focused exercises has the effects on Time to Stabilization after Anterior Cruciate Ligament Reconstruction". The purpose of these study to determine the relationship between muscle strength and time taking to increase the performance of knee. The main findings suggesting that rehabilitation program targets on strengthen the hip muscles in comparison with traditional exercises of knee demonstrate an improvement of knee functions in individual with Anterior cruciate ligament reconstruction (ACLR).

In previous studies there is very less literature regarding determining effects of the clamshells exercises on extension lag after anterior cruciate ligament reconstruction. Therefore there is a dire need to explore the effect of the clamshells exercises on post anterior cruciate ligament reconstruction extension lag. This study aims in the management of pain disability and functional impairment in persons with extension lag with clamshells exercises after ACL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* Both Genders (male & female)
* History of Anterior Cruciate Ligament Reconstruction (ACLR) between 1-3 years

Exclusion Criteria:

* Any other previously serious knee pain and/or surgery.
* Limiting of knee range of motion.
* Any traumatic conditions around the knee, or any infectious or tumors conditions
* Pregnancy, any recently underwent abdominal and back surgery.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
extension knee range of motion | 4th week
  Change from the baseline ROM of knee extension was taken with the help of goniomter

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Imran, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No